CLINICAL TRIAL: NCT06092034
Title: Gene Therapy for Danon Disease: A Phase 2 Study Evaluating the Efficacy and Safety of Intravenously Administered Adeno-Associated Virus Serotype 9 (rAAV9) Vector Containing the Human LAMP2 Isoform B Transgene (RP-A501; AAV9.LAMP2B) in Male Patients With Danon Disease
Brief Title: A Gene Therapy Study of RP-A501 in Male Patients With Danon Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rocket Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP-A501-0123
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Danon Disease
Keywords: Hypertrophic Cardiomyopathy; HCM; X-linked disease; LAMP2; Pediatric; Skeletal Myopathies; Cardiomyopathy; Lysosomal Storage Disorder; Left Ventricular Hypertrophy
MeSH Terms: conditions — Glycogen Storage Disease Type IIb; Cardiomyopathy, Hypertrophic; Cardiomyopathies; Lysosomal Storage Diseases; Hypertrophy, Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RP-A501 (Experimental): One planned dose of RP-A501 in cohorts of subjects with a confirmed diagnosis of Danon Disease.
  Interventions: Genetic: RP-A501

INTERVENTIONS:
Genetic: RP-A501 — RP-A501 is a gene therapy product consisting of a rAAV9 capsid containing the human LAMP2B transgene which will be administered as a single IV infusion.

SUMMARY:
This is a single arm Phase 2 trial to evaluate the efficacy and safety of RP-A501, a recombinant adeno-associated virus serotype 9 (AAV9) containing the human lysosome-associated membrane protein 2 isoform B (LAMP2B) transgene, in male patients with Danon Disease.

DETAILED DESCRIPTION:
The study is a single arm Phase 2 clinical trial to characterize the safety and efficacy of RP-A501, a recombinant adeno-associated serotype 9 (rAAV9 capsid containing the human lysosome-associated membrane protein 2 isoform B (LAMP2B) transgene) in male patients with Danon Disease.

Male subjects ≥8 years of age will receive a single intravenous infusion of RP-A501.

ELIGIBILITY:
Key Inclusion Criteria:

1. Documentation of a pathogenic or likely pathogenic variant of the LAMP2 gene.
2. Male.
3. Age ≥8 years.
4. Evidence of left ventricular hypertrophy with preserved systolic function phenotype as defined by each of the following:

   1. Abnormal thickening of Left ventricular wall,
   2. Left ventricular ejection fraction (LVEF) ≥ 50%.
5. New York Heart Association (NYHA) Class II to III.
6. High sensitivity Troponin I (hsTnI) ≥20% above the upper limit of normal (ULN)
7. Ability to comply with study procedures including investigational therapy and follow-up evaluations.

Key Exclusion Criteria:

1. Anti-AAV9 neutralizing antibody titer >1:40.
2. Severe heart failure or requirement for advanced therapies.
3. History of intracardiac thrombosis or arterial thromboembolic events including stroke, transient ischemic attack (TIA), acute coronary syndrome, myocardial infarction or unstable angina.
4. Prior cardiac or other organ (lung, liver, other) transplantation.

Min Age: 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy via primary endpoint comprised of LAMP2 myocardial tissue expression and left ventricular mass index | 12 Months post-infusion
  Increase of myocardial tissue expression of LAMP2 protein and decrease in left ventricular mass index (LVMI).

SECONDARY OUTCOMES:
Evaluation of efficacy via components of the primary endpoint - LAMP2 | 12 months post infusion
  Increase in LAMP2 protein expression
Evaluation of efficacy via components of the primary endpoint - Left Ventricular Mass Index (LVMI) | 12 months post infusion
  Decrease in Left Ventricular Mass Index (LVMI)
Evaluation of efficacy via biomarker evidence of myocardial injury - High Sensitivity Troponin I (hsTnI) | 12 months post infusion
  Decrease in high sensitivity Troponin I (hsTnI)
Evaluation of efficacy via biomarker evidence of myocardial injury - N-Terminal Prohormone of Brain Natriuretic Peptide (NT-proBNP) | 12 months post infusion
  Decrease in N-terminal prohormone of brain natriuretic peptide (NT-proBNP)
Evaluation of efficacy via assessment of event-free survival | 60 months post infusion
  1. Event free survival with events defined as death, heart transplant, mechanical circulatory support (MCS) or heart failure hospitalization
  2. Incidence of death, heart transplant, MCS, or heart failure hospitalization
Evaluation of safety | 60 months post infusion
  Incidence, severity and duration of treatment emergent safety events.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rossano, MD, Principal Investigator — Children's Hospital of Philadelphia; Barry Greenberg, MD, Principal Investigator — University of California, San Diego
Locations (6):
- United States (3):
  - University of California, San Diego, La Jolla, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- German Heart Center Munich, Munich, Germany
- Meyer Childrens Hospital, Florence, Italy
- Great Ormund Street Hospital & UCL Institute of Cardiovascular Science, London, United Kingdom